CLINICAL TRIAL: NCT03912298
Title: Effect of Opioid Taper on Pain Responses in Patients With Chronic Pain
Brief Title: Opioid Taper Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 831447; 1R21DA046364-01A1 (NIH)
Record Dates: First submitted 2019-04-04; First posted 2019-04-11 (Actual); Results first posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Opioid Taper Pain perception — Pain Responses: The primary dependent variable, pain, will be measured using two highly reliable and valid pain induction techniques, the CPT and QST, employing procedures consistent with those described in the literature. Order of pain testing will vary, and three aspects of the pain response will be captured at each study session: evoked pain; temporal summation; and conditioned pain modulation, which map on to the hypothesized peripheral, spinal and supra-spinal mechanisms of OIH. Protocols for each assay have been uploaded.

SUMMARY:
The purpose of this study is to determine the effect of opioid taper on pain sensitivity in patients with chronic pain. In a well-characterized sample of men and women with chronic neuropathic pain on high-dose opioid therapy, experimental pain responses (cold-pressor, quantitative sensory testing) will be serially described over the course of and following an individualized opioid taper. In addition, functional improvements and subject-level predictors of response will be described.

DETAILED DESCRIPTION:
The overall Specific Aim of this proposal is to determine the effect of opioid taper on pain sensitivity in patients with chronic pain. Specifically, in a well-characterized sample of men and women with chronic neuropathic pain and receiving high-dose opioid therapy (>100mg morphine equivalents/day [MED]), experimental pain responses will be serially described over the course of an individualized opioid taper to a safer dose of 90mg MED for up to 12 months. Changes will be inspected within-subject over time, and pain perception will be measured with two valid and reliable experimental pain induction techniques commonly used to measure OIH (cold-pressor, quantitative sensory testing); in addition, related functional improvements and subject-level predictors of response will be described.

Hypothesis 1. Subjects undergoing opioid taper will have improved pain responses over time compared to within-subject baseline as measured by cold-pressor and quantitative sensory pain testing.

Hypothesis 2. Improvements in experimental pain responses will be positively related to improved functional outcomes compared to within-subject baseline as measured by the PROMIS physical, mental and social health measures.

Hypothesis 3. Degree of improvement in experimental pain responses related to opioid taper will be predicted by demographic, pain, and opioid use history characteristics of the subject.

Data showing that pain perception improves as opioids are withdrawn would provide an evidence-based, mechanistic rationale for opioid taper in patients with chronic pain and have the potential to support a sea-change in opioid prescription practices. In that ongoing opioid therapy brings with it significant health risks for the patient and the community, it is critical that empirical evidence of its efficacy be demonstrated to balance the benefits with the risks of adverse events, potential misuse and abuse, and patient safety.

ELIGIBILITY:
Inclusion Criteria:

1. between ages of 21-70;
2. documented chronic neuropathic non-malignant pain condition of at least one year duration;
3. on >100mg/day MED for at least 6 months;
4. have fully engaged in all prescribed non-opioid pain management treatments;
5. willing to undergo prescribed opioid taper;
6. otherwise in good physical and mental health, or in the care of a physician who is willing to take responsibility for such treatment;
7. able to understand the purpose and instructions of the study, and provide informed consent as approved by the University of Pennsylvania IRB.

Exclusion Criteria:

1. meet diagnostic criteria for an active substance use disorder other than nicotine;
2. be acutely psychotic, severely depressed, and/or in need of inpatient psychiatric treatment,
3. have a neurological or psychiatric illness that would affect pain responses, including anxiety disorders;
4. have a history of heart disease, stroke, or a pacemaker or uncontrolled high blood pressure. Good cardiovascular health is stipulated to ensure subjects can tolerate the sympathetic nervous system responses associated with the pain induction procedures.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will consist of 25 male and female adults with chronic neuropathic pain on opioid therapy and preparing to voluntarily undergo a prescribed opioid taper.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Compton, RN, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Pain Medicine Center Tuttleman Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dowell D, Haegerich TM. Changing the Conversation About Opioid Tapering. Ann Intern Med. 2017 Aug 1;167(3):208-209. doi: 10.7326/M17-1402. Epub 2017 Jul 11. No abstract available. PMID 28715842
- [Background] Peles E, Schreiber S, Hetzroni T, Adelson M, Defrin R. The differential effect of methadone dose and of chronic pain on pain perception of former heroin addicts receiving methadone maintenance treatment. J Pain. 2011 Jan;12(1):41-50. doi: 10.1016/j.jpain.2010.04.009. Epub 2010 Jun 19. PMID 20561825
- [Background] Wang H, Fischer C, Chen G, Weinsheimer N, Gantz S, Schiltenwolf M. Does long-term opioid therapy reduce pain sensitivity of patients with chronic low back pain? Evidence from quantitative sensory testing. Pain Physician. 2012 Jul;15(3 Suppl):ES135-43. PMID 22786452
- [Derived] Compton P, Halabicky OM, Aryal S, Badiola I. Opioid Taper is Associated with Improved Experimental Pain Tolerance in Patients with Chronic Pain: An Observational Study. Pain Ther. 2022 Mar;11(1):303-313. doi: 10.1007/s40122-021-00348-8. Epub 2022 Jan 12. PMID 35020185

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Pain Patients Undergoing Opioid Taper: Chronic pain patients undergoing an individualized opioid taper to a safer daily dose of opioid for up to one year.
Period: Overall Study
Arm/Group | Chronic Pain Patients Undergoing Opioid Taper
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Chronic Pain Patients Undergoing Opioid Taper: Chronic pain patients undergoing opioid taper
Arm/Group | Chronic Pain Patients Undergoing Opioid Taper
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 6
  Race: Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
mg morphine equivalents/day or MME/day [Mean (Standard Deviation); unit: daily morphine mg equivalents] | 291.85 (182.62)

OUTCOME MEASURES:

1. Primary Outcome: Pain Perception Measured Using the Cold-pressor Test (CPT)
Description: Pain perception will be measured using the cold-pressor test (CPT) employing procedures consistent with those described in the literature. Order of pain testing will vary, and three aspects of the pain response will be captured at each study session: evoked pain; temporal summation; and conditioned pain modulation, which map on to the hypothesized peripheral, spinal and supra-spinal mechanisms of OIH. Reported are cold-pressor pain tolerance prior to and following taper.
Time Frame: up to one year (length of taper individualized and varies)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Chronic Pain Patients Undergoing Opioid Taper
Number analyzed (Participants) | 7
seconds
  pre taper pain tolerance (baseline) | 24.01 (20.63)
  post-taper pain tolerance (timeframe variable) | 42.02 (41.83)

2. Primary Outcome: Conditioned Pain Modulation Measured Using the Quantitative Sensory Testing (QST)
Description: Conditioned pain modulation will be measured using the quantitative sensory testing (QST) employing procedures consistent with those described in the literature to capture supra-spinal mechanisms of OIH. To detect conditioned modulation, the subject is asked to verbally report the severity of pain experienced on a visual analogue scale (0- no pain, 10-worst pain ever) to a three-second painful heat stimulus (47○C) delivered at 12-15 second intervals, in the presence or absence of the non-dominant limb being immerged in a cold-water bath (12○C). The reported value is the difference between the average of pain scores reported in the absence of vs. the presence of the counter-stimulation. Reported are changes in the conditioned pain modulation assay both prior to and following taper. Taper is individualized thus length of taper varies between subjects.
Time Frame: up to one year (individualized, variable taper length)
Measure: Mean (Standard Deviation); unit: units on a visual analogue scale
Arm/Group | Chronic Pain Patients Undergoing Opioid Taper
Number analyzed (Participants) | 7
units on a visual analogue scale
  pre-taper conditioned pain modulation (baseline) | -0.14 (0.42)
  post taper conditioned pain modulation (individualized taper, thus time length varies) | -0.40 (0.79)

ADVERSE EVENTS:
Time Frame: up to 12 months
Description: Subjects were carefully screened and excluded from participation if they had any risk factors putting them at risk for serious adverse events and mortality. Presence of adverse event s assessed on a biweekly basis.
Arm/Group | Chronic Pain Patients Undergoing Opioid Taper
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT03912298/Prot_SAP_000.pdf